CLINICAL TRIAL: NCT06613100
Title: A Phase 1b, Open-Label, Multicenter Study Evaluating the Safety, Tolerability, and Feasibility of Neoadjuvant Xaluritamig Therapy Prior to Radical Prostatectomy in Subjects With Newly Diagnosed Localized Intermediate or High-Risk Prostate Cancer
Brief Title: Evaluation of Neoadjuvant Xaluritamig in Localized Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230237; 2024-511965-13 (Other: EU CT Number)
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: Xaluritamig; AMG509; Localized Prostate Cancer; Prostate Cancer; Neoadjuvant Therapy; Immunotherapy; T-Cell Engager; STEAP1
MeSH Terms: conditions — Prostatic Neoplasms | interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A - Xaluritamig (Experimental): Xaluritamig will be administered prior to radical prostatectomy.
  Interventions: Drug: Xaluritamig
- Cohort B - Xaluritamig with an Oral GnRH Antagonist (Experimental): Xaluritamig will be administered prior to radical prostatectomy. Participants will also receive an oral GnRH antagonist continuously up to the time of planned radical prostatectomy.
  Interventions: Drug: Xaluritamig; Drug: GnRH Antagonist

INTERVENTIONS:
Drug: Xaluritamig — Intravenous (IV) infusion
  Other Names: AMG 509
Drug: GnRH Antagonist — Oral administration
  Arms: Cohort B - Xaluritamig with an Oral GnRH Antagonist

SUMMARY:
The primary objectives of this study are to evaluate the safety and tolerability of xaluritamig administered as monotherapy or in combination with an oral Gonadotropin-releasing Hormone (GnRH) antagonist in the neoadjuvant setting followed by radical prostatectomy, and to evaluate the feasibility and safety of a radical prostatectomy following xaluritamig administered as monotherapy or in combination with an oral GnRH antagonist in the neoadjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all the following criteria apply:

* Participants planned to undergo radical prostatectomy.
* Histologically or cytologically confirmed adenocarcinoma of the prostate at initial biopsy, without neuroendocrine differentiation, signet cell, or small cell features. Intermediate- or high-risk localized prostate cancer, defined as:

  * Gleason score of 4+3 or higher AND initial PSA (iPSA) >10 OR
  * Clinically advanced (cT3) on Magnetic Resonance Imaging (MRI) obtained within 3 months prior to screening AND/OR
  * Positive locoregional lymph nodes as detected by prostate-specific membrane antigen-positron emission tomography (PSMA-PET) scans OR ≤ 5 local lymph nodes on MRI can be enrolled.
* Participants must have undergone a PSMA-PET (CT or MRI) scan within 3 months prior to screening as part of the standard of care (SOC).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Prior treatment for participant's prostate cancer.

  - Exception: Participants intended for enrollment in cohort B may have received an oral GnRH antagonist up to 3 months prior to the start of screening.
* Any evidence of metastases outside of the surgical resection field identified by conventional imaging or PSMA-PET scans.
* Confirmed history or current autoimmune disease or other diseases resulting in permanent immunosuppression or requiring permanent immunosuppressive therapy.
* Participants with symptoms and/or clinical signs and/or radiographic signs that indicate an acute and/or uncontrolled active systemic infection within 7 days prior to the first dose of study treatment:

  - Participant has known active infection requiring antibiotic treatment. Upon completion of antibiotics and resolution of symptoms, the participant may be considered eligible for the study from an infection standpoint.
* Recent history of arterial or venous thrombosis (eg, stroke, transient ischemic attack, pulmonary embolism, or deep vein thrombosis) within 6 and 3 months prior to the first dose of study treatment, respectively. Note: Participants with a history of venous thrombosis must be on stable anti-coagulation.
* Myocardial infarction and/or symptomatic congestive heart failure (New York Heart Association ≥ class II) within 12 months of first dose of xaluritamig with the exception of ischemia or non-ST segment elevation myocardial infarction controlled with stent placement more than 6 months prior to first dose of xaluritamig.
* Requirement for chronic systemic corticosteroid therapy unless stopped (with adequate tapering) within 7 days prior to dosing.
* Currently receiving treatment in another investigational device or drug study, or less than 4 weeks (since ending treatment on another investigational device or drug study[ies]). Other investigational procedures and participation in observational research studies while participating in this study are excluded with the exception of investigational scans.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2027-01-22 (Estimated); Study Completion 2030-01-23 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Experienced Treatment-emergent Adverse Events | Up to 45 months
  Inclusive of adverse events, serious adverse events, and changes in vital signs and clinical laboratory tests.
Number of Participants who Experienced Treatment-related Adverse Events | Up to 28 months
Number of Participants who Received Radical Prostatectomy After Completing Xaluritamig Treatment | Up to 25 months
Number of Participants who Experienced Complications of Radical Prostatectomy According to Clavien-Dindo Classification | Up to 28 months

SECONDARY OUTCOMES:
Change in Prostate-specific Antigen (PSA) Levels from Baseline to End of Xaluritamig Treatment | Up to 25 months
Prostate Imaging-Reporting and Data System (PI-RADS) Score | Up to 25 months
Pathological Complete Response (pCR) Following Radical Prostatectomy | Up to 25 months
Minimal Residual Disease (MRD) | Up to 25 months
Number of Participants who Rise to PSA ≥ 0.2 ng/mL Post-radical Prostatectomy | Up to 45 months
Time to PSA Rise ≥ 0.2 ng/mL Post-radical Prostatectomy | Up to 45 months
Undetectable PSA at SFU | Up to 26 months
PSA Progression-free Survival | Up to 45 months
Maximum Serum Concentration (Cmax) of Xaluritamig | Up to 45 months
Time to Maximum Concentration (Tmax) of Xaluritamig | Up to 45 months
Area Under the Concentration Time Curve (AUC) Over the Dosing Interval | Up to 45 months
Accumulation Following Multiple Dosing | Up to 45 months
Half-life (t1/2) of Xaluritamig | Up to 45 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (8):
- United States (6):
  - University of California San Francisco, San Francisco, California
  - Washington University, St Louis, Missouri
  - The Ohio State University, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Germany (2):
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com